CLINICAL TRIAL: NCT00307008
Title: An Open, Phase II Study to Evaluate the Response Rate to the Licensed Single-Dose Polysaccharide Pneumococcal Vaccine Pneumovax 23™ (MSD Aventis Pasteur) in Elderly Population.
Brief Title: Study to Evaluate the Response Rate to the Licensed Pneumovax 23™ in Elderly Population.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 513026/004; 100421; 100436
Record Dates: First submitted 2006-03-24; First posted 2006-03-27 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2011-09

CONDITIONS: Streptococcus Pneumoniae Vaccines
Keywords: Prophylaxis Invasive pneumococcal diseases and pneumonia
MeSH Terms: conditions — Pneumonia | interventions — 23-valent pneumococcal capsular polysaccharide vaccine

ARMS (1):
- Group A (Experimental)
  Interventions: Biological: Pneumovax 23™

INTERVENTIONS:
Biological: Pneumovax 23™ — Single dose intramuscular injection

SUMMARY:
Streptococcus pneumoniae are bacteria which normally live in the upper respiratory tract of humans. However, these bacteria can also cause severe infectious diseases such as pneumonia, septicemia and meningitis. Elderly subjects are especially vulnerable to these infections, and the diseases can result in death. The currently available licensed Streptococcus pneumoniae vaccine is recommended for prevention of pneumococcal diseases in individuals over the age of 65. However, the antibody level elicited by this vaccine, is not always satisfactory in elderly people. To overcome the problem, GlaxoSmithKline Biologicals is currently developing candidate vaccines that are hoped to work better than the currently available vaccines. As a first step in this development, the present study is being conducted in order to evaluate the immune response to the currently marketed vaccine.

DETAILED DESCRIPTION:
Since influenza vaccination is recommended in the age range of the study population, Fluarix™ (GlaxoSmithKline Biologicals) vaccine will be offered free of charge for the study period (3 consecutive years), to be used by Investigators according to national vaccination schedule/practice.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007

ELIGIBILITY:
Inclusion criteria

* Subjects who the investigator believes will comply with the requirements of the protocol.
* A male or female >= 65 years at the time of the first vaccination.
* Written informed consent obtained from the subject.

Exclusion criteria

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period or participation to another pharmaceutical/vaccine study.
* Previous vaccination against Streptococcus pneumoniae.
* History of administration of an experimental vaccine containing MPL or QS21.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Planned administration of a vaccine not foreseen by the study protocol within 2 weeks before and after first dose of vaccines, excluding influenza vaccine which can be administered at any time, including co-administration with Pneumovax23™.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* Current serious neurologic or mental disorders.
* Inflammatory processes such as known chronic active infections (e.g.Hep B, C).
* All malignancies (excluding non-melanic skin cancer) and lymphoproliferative disorders diagnosed or treated actively during the past 5 years.
* Acute disease at the time of enrolment.
* Chronic disease that might preclude participation to the whole study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1198 (Actual)
Dates: Start 2003-10; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Response rate to 11 vaccine serotypes | One month post vaccination

SECONDARY OUTCOMES:
Anti-polysaccharide total IgG ELISA for 11 vaccine pneumococcal serotypes | At all time points
Opsonophagocytic activity against 11 vaccine pneumococcal serotypes in a subset of subjects | At Day 0 and Day 30.
The rank of subjects from "poorest responder" to "best responder" based on the number of serotypes each subject responds to | One month post vaccination
Persistence of the immune response in a subset of subjects. | Until Month 36.
Opsonophagocytic activity response in a subset of subjects. | At Day 30
Occurrence of serious adverse events (SAE). | Up to 1 month after vaccination.
Occurrence of study related SAEs. | Throughout the study period.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Sweden (5):
  - GSK Investigational Site, Eskilstuna
  - GSK Investigational Site, Jönköping
  - GSK Investigational Site, Skövde
  - GSK Investigational Site, Uppsala
  - GSK Investigational Site, Västerås